CLINICAL TRIAL: NCT03392766
Title: Comparison of Fiberoptic Intubation Between Double Lumen Tube and Single Lumen Tube in Patients With Semi-rigid Neck Collar Immobilization of the Cervical Spine.
Brief Title: Fiberoptic Bronchoscope of Double Lumen Tube and Single Lumen Tube in Patients With Semi-regid Neck Collar.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, DAE HEE KIM, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AJIRB-DEV-OBS-17-247
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Intubation;Difficult; Thoracic Diseases
Keywords: fibreoptic intubation; double lumen tube; difficult intubation
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single lumen tube and bronchial blocker (Experimental): neck collar apply. fibreoptic intubation with single lumen tube and brochial blocker
  Interventions: Device: single lumen tube and bronchial blocker
- Double lumen tube (Experimental): neck collar apply. fibreoptic intubation with double lumen tube
  Interventions: Device: double lumen tube

INTERVENTIONS:
Device: single lumen tube and bronchial blocker — neck collar apply. fibreoptic intubation with single lumen tube and bronchial blocker.
  Arms: Single lumen tube and bronchial blocker
Device: double lumen tube — neck collar apply. fibreoptic intubation with double lumen tube.
  Arms: Double lumen tube

SUMMARY:
Many intrathoracic procedures demand optimal collapse of the operative lung to facilitate surgical exposure. Single-lung ventilation can be achieved using a double-lumen tube (DLT), a Univent tube, or an independent bronchial blocker. Insertion of a DLT using a direct laryngoscope can be more difficult than that of single-lumen tube (SLT), especially in patients for whom airway difficulty is anticipated. The safest of the proposed methods involves the placement of an SLT with the aid of an fibreoptic bronchoscope (FOB), following which the SLT is replaced with a DLT using an airway exchange technique in these patients. HumanBroncho® (Insung Medical, Seoul, Korea) is a new silicone DLT with a soft, flexible, non-bevelled, wire-reinforced tip. The oval shape, obtuse angle, and short lateral internal diameter of the bronchial lumen and its flexibility may allow for advancement to the trachea over the FOB with as much as ease as a standard SLT. In the present study, the investigators aimed to test the hypothesis that the HumanBroncho® DLT would be non-inferior to a standard SLT with regard to intubation time over an FOB in patients with semi-rigid neck collar simulating difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery requiring one lung ventilation. American Society of Anesthesiologist, Physical Status 1,2

Exclusion Criteria:

* abnormality of upper airway gastroesophageal disease risk of aspiration BMI > 35

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
intubation time | through study completion, an average of 4 hour
  the time from the passage of the fibreoptic bronchoscope beyond the teeth, to tracheal tube positioning above the carina.

SECONDARY OUTCOMES:
insertion time | through study completion, an average of 4 hour
  the time from the passage of the fibreoptic bronchoscope beyond the teeth, to fibreoptic bronchoscope positioning above the carina
railroading time | through study completion, an average of 4 hour
  the time from fibreoptic bronchoscope positioning above the carina to tracheal tube positioning above the carina.
grade of ease of insertion over fibreoptic bronchoscope | through study completion, an average of 4 hour
  1, no difficulty passing the tube; 2, obstruction while passing the tube, relieved by withdrawal and a 90° counter-clockwise rotation; 3, obstruction necessitating more than one manipulation or external laryngeal manipulation; 4, direct laryngoscopy was required.
trauma around the glottis | through study completion, an average of 4 hour
  fibreoptic observation of the glottic bleeding.
complication at the post-anesthesia care unit | through study completion, an average of 4 hour
  hoarseness, sore throat, swallowing difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hee Kim, M.D., Principal Investigator — Ajou unversity hospital
Locations (1):
- Ajou universiry hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang S, Chae YJ, Kim DH, Bae SY, Yoo JY. Comparison of silicone double-lumen tube and polyvinyl chloride single-lumen tube in fiberoptic tracheal intubation on a difficult airway model: a randomized controlled non-inferiority trial. Sci Rep. 2023 May 24;13(1):8397. doi: 10.1038/s41598-023-35635-1. PMID 37225777